CLINICAL TRIAL: NCT06454214
Title: 3D Structural Imaging of Human Breast Tissues
Status: Not yet recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202405097RINB
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Human Breast Tissues
Keywords: breast tumor; tumor assessment; tumor microenvironment; digital pathology; 3D pathology
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control breast tissues (normal breast tissues): Normal tissue contained within the surgically excised specimen
  Interventions: Device: Multi-photon microscopy
- Cancerous breast tissues: Tumor tissue contained within the surgically excised specimen
  Interventions: Device: Multi-photon microscopy

INTERVENTIONS:
Device: Multi-photon microscopy — To conduct 3D structural imaging on human breast tissues

SUMMARY:
This project aims to develop an advanced ex vivo medical microscopic imaging technology. By developing breast tissue staining techniques, acquiring microscopic images, and performing structural reconstruction, we seek to observe the 3D structure of breast tissue. This includes examining cell distribution, mammary ducts, and blood vessel distribution, to explore the different biological characteristics between normal breast tissue and various types of cancerous tissues.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and above.
* Patients clinically diagnosed with breast cancer.

Exclusion Criteria:

* Patients unable to provide consent (e.g., inability to speak, inability to communicate in Chinese, etc.).
* Patients for whom a definitive pathological diagnosis cannot be established.
* Patients suitable only for biopsy and not for surgical excision.
* Excised tissue showing severe radiation-induced changes under pathological examination.
* Tumor specimens smaller than 1 cm.
* Patients with ductal carcinoma in situ (DCIS).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This research project aims to recruit 100 subjects and acquire three-dimensional images of the breast tissues. After reconstructing these images, the study will explore the diverse three-dimensional structures of tumor tissues and compare them with the structures of normal breast tissues.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-06-04 (Estimated); Study Completion 2027-06-04 (Estimated)

PRIMARY OUTCOMES:
Accuracy dependency on staining dye selection | 3 years
  Using other types of staining agents, compare the diagnostic accuracy of the results with those of traditional pathological staining agents.

SECONDARY OUTCOMES:
Comparison between 3D pathology vs. FFPE on breast cancer samples with a focus on image contrast | 3 years
  Verify whether the contrast and other conditions can provide pathologists with critical information for interpretation. The images will also be compared with the results observed using traditional pathology methods.

IPD SHARING:
Plan to Share IPD: No
This study will not share individual participant data.